CLINICAL TRIAL: NCT01001754
Title: Randomized, Controlled Phase 2a/b Study of the Efficacy and Safety of PEG-rIL-29 Administered in Combination With Ribavirin to Treatment-Naive Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Efficacy and Safety Study of PEG-rIL-29 Plus Ribavirin to Treat Chronic Hepatitis C Virus Infection
Acronym: EMERGE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ZymoGenetics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 526H04; 2009-011786-80 (EudraCT Number)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Hepatitis C, Chronic; PEGylated recombinant interleukin 29; PEG-interferon lambda; Interleukin 29; Virus; Infection; Liver Diseases
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Virus Diseases; Infections; Liver Diseases | interventions — peginterferon lambda-1a; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PEG-rIL-29 at 120 µg (Experimental)
  Interventions: Drug: PEG-rIL-29; Drug: Ribavirin
- PEG-rIL-29 at 180 µg (Experimental)
  Interventions: Drug: PEG-rIL-29; Drug: Ribavirin
- Peginterferon alfa-2a at 180 µg (Active Comparator)
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: PEG-rIL-29 — Weekly SC injections in combination with ribavirin for up to 48 weeks
  Arms: PEG-rIL-29 at 120 µg; PEG-rIL-29 at 180 µg
Drug: Peginterferon alfa-2a — Weekly SC injections in combination with ribavirin for up to 48 weeks
  Other Names: PEGASYS
  Arms: Peginterferon alfa-2a at 180 µg
Drug: Ribavirin — Daily oral administration (400-600 mg BID)

SUMMARY:
Interleukin 29 (IL-29) is a substance that is produced in the body to help fight viral infections. The purpose of this study is to evaluate the safety and antiviral effects of several different doses of PEG-rIL-29 (a man-made form of IL-29) when it is given in combination with daily oral doses of ribavirin (an antiviral drug) to subjects with hepatitis C infection who have received no prior treatment for this disease.

DETAILED DESCRIPTION:
PEG-rIL-29 (also known as PEG-interferon lambda) is a unique Type III interferon molecule that has demonstrated antiviral activity when administered weekly for 4 weeks to treatment-relapsed and treatment-naive subjects with genotype 1 hepatitis C virus (HCV) infection. Because PEG-rIL-29 binds to a unique receptor with a more limited distribution than the receptor for interferon (IFN)-α, it may have the potential to treat HCV without some of the treatment-limiting side effects associated with IFN-α-based therapies. The purpose of this Phase 2a/b randomized, controlled, multicenter study is to compare the safety and efficacy of PEG-rIL-29 and peginterferon alfa-2a, both administered subcutaneously weekly for up to 48 weeks in combination with daily oral ribavirin, in treatment-naive subjects with chronic genotype 1, 2, 3, or 4 HCV infection. The initial part of the study (Phase 2a) will be conducted as an open-label study; the second part of the study (Phase 2b) will be conducted as a blinded study. The above information provided in this listing is specific to the Phase 2b portion of the study. In addition, two small open-label substudies will be conducted to evaluate the efficacy of 24-week treatment with PEG-rIL-29 and ribavirin in subjects with HCV genotype 1 who have a particular genetic polymorphism associated with favorable response (n=60) and to evaluate the efficacy of 16-week treatment with PEG-rIL-29 and ribavirin in subjects with HCV genotype 2 or 3 (n=30).

ELIGIBILITY:
Inclusion Criteria:

* No prior therapy for chronic HCV, other than up to 2 weeks of single-agent therapy with a direct-acting antiviral agent, including but not limited to, a protease or polymerase inhibitor
* HCV genotype 1, 2, 3, or 4
* HCV RNA ≥100,000 IU/mL
* ALT and AST ≤5.0 × ULN
* Documented absence of cirrhosis
* Able to comprehend the investigational nature of this study and sign an informed consent form

Exclusion Criteria:

* Mixed genotype HCV infection
* Current or prior history of decompensated liver disease
* Received any investigational drug, including a direct-acting antiviral agent, within 60 days prior to receiving study drug
* Positive test for hepatitis B surface antigen, human immunodeficiency virus (HIV)-1, or HIV2 antibody at screening
* Active substance abuse, such as alcohol, or inhaled or injected drugs, within 6 months

Additional inclusion and exclusion criteria are specified in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
HCV RNA | At week 12, week 24, or week 48
Incidence and severity of adverse events | Through week 12, week 40, or week 48

SECONDARY OUTCOMES:
Incidence and severity of adverse events and laboratory abnormalities | Up to week 72
HCV RNA | Up to week 72
PD biomarkers | Up to week 72
Quality of life assessments | Up to week 72
Serum drug concentration profile | Up to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hillson, MD, Study Director — ZymoGenetics
Locations (79):
- United States (29):
  - Beverly Hills, California
  - Coronado, California
  - La Jolla, California
  - Palm Springs, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Lutherville, Maryland
  - Detroit, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Manhasset, New York
  - New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Statesville, North Carolina
  - Philadelphia, Pennsylvania
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Newport News, Virginia
  - Seattle, Washington
- Australia (13):
  - Herston, Queensland
  - Adelaide
  - Camperdown
  - Clayton
  - Fitzroy
  - Fremantle
  - Greenslopes
  - Herston
  - Kogarah
  - Melbourne
  - Penrith
  - Perth
  - Westmead
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Canada (3):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
- France (2):
  - Paris
  - Pessac
- Germany (13):
  - Bochum
  - Cologne
  - Düsseldorf
  - Essen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Göttingen
  - Hamburg
  - Hanover
  - Heidelberg
  - Mainz
  - München
  - Tübingen
- Milan, Italy
- Poland (5):
  - Bialystok
  - Krakow
  - Racibórz
  - Wroclaw
  - Łańcut
- Santurce, Puerto Rico
- Romania (3):
  - Bucharest
  - Iași
  - Timișoara
- Spain (5):
  - Barcelona
  - Madrid
  - Majadahonda
  - Seville
  - Valencia

REFERENCES:
- [Derived] Wang X, Hruska M, Chan P, Ahmad A, Freeman J, Horga MA, Hillson J, Kansra V, Lopez-Talavera JC. Derivation of Phase 3 dosing for peginterferon lambda-1a in chronic hepatitis C, Part 1: Modeling optimal treatment duration and sustained virologic response rates. J Clin Pharmacol. 2015 Jan;55(1):63-72. doi: 10.1002/jcph.363. Epub 2014 Jul 24. PMID 25043197
- [Derived] Hruska M, Wang X, Chan P, Ahmad A, Freeman J, Horga MA, Hillson J, Kansra V, Lopez-Talavera JC. Derivation of Phase 3 dosing for peginterferon lambda-1a in chronic hepatitis C, Part 2: Exposure-response analyses for efficacy and safety variables. J Clin Pharmacol. 2015 Jan;55(1):73-80. doi: 10.1002/jcph.361. Epub 2014 Jul 24. PMID 25042797